CLINICAL TRIAL: NCT05219344
Title: Effects of Different Volumes of Tissue Flossing Around Thigh Muscle on Neuromuscular Function
Brief Title: Tissue Flossing and Lower Limb Neuromuscular Function
Acronym: MF2-TMG-CMJ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ljubljana (Other)
Responsible Party: Principal Investigator, Armin Paravlic, Faculty of Sport, University of Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Thigh Flossing 2022
Record Dates: First submitted 2022-01-20; First posted 2022-02-02 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Physical Performance; Neuromuscular Function; Tissue Flossing; Ischemic Preconditioning
Keywords: Physical Performance, Neuromuscular Function, CMJ, TMG, PAP
MeSH Terms: interventions — Ischemic Preconditioning

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The kinesiologist (care provider), investigator and assessors will be blind for group allocation of the participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One set of muscle flossing (Experimental): This group will receive one set of muscle flossing around the thigh with low pressure. Pressure will be individualized based on thigh circumferences.
  Interventions: Procedure: Tissue flossing
- Two sets of muscle flossing (Active Comparator): This group will receive two sets of muscle flossing around the thigh with low pressure. Pressure will be individualized based on thigh circumferences.
  Interventions: Procedure: Tissue flossing

INTERVENTIONS:
Procedure: Tissue flossing — After the standardized warm-up, participants will be instructed to stand still with their legs shoulder-width apart. The floss band (1.3 mm thick, 50 mm wide, 2 meters long, and strength level 3), consisting of a thick elastic latex band (COMPRE Floss, Sanctband), will be applied bilaterally around the distal third of the thigh. The applied pressure will be individualized by thigh circumferences, whereas low target pressure was chosen for this study, showing potential to elicit the most beneficial outcomes following flossing. The pressure will be monitored by the PicoPress device, which was placed at the middle distance of the application of the floss band to ensure that the entire surface of the pressure sensors was always completely covered. The flossing will be applied for 2 minutes with 2 minutes rest between sets. During flossing application subjects will be instructed to conduct 10 deep squats followed by 15 repetitions of knee extensions without added weight.
  Other Names: ischemic preconditioning

SUMMARY:
There is no study investigating different volumes, that is various sets of the configuration of tissue flossing on neuromuscular function. Previously, investigators found that 3 sets of TF impaired neuromuscular function assessed with TMG. Therefore, the aim is to compare the effects of one and two sets of TS on countermovement jump (CMJ) performance and muscle contractile properties.

DETAILED DESCRIPTION:
The primary purpose of the study will be to examine the differences in one and two sets of applying tissue flossing to the thigh muscles on neuromuscular function using tensiomyography (TMG) and CMJ, while considering several measurement points after flossing application (i.e., +0.5min, +3min, +6min, +9min, +12min, +15min). A better understanding of the effects of flossing on acute performance enhancement as well as on individual muscle contractile properties could help practitioners to develop specific pre-conditioning activities and consequently improve athletic performance on the field. The investigators hypothesized that: (i) the application of tissue flossing will improve the contraction time of the vastus lateralis muscle as well as the maximal jumping performance, regardless of sets of configuration.

ELIGIBILITY:
Inclusion Criteria:

* healthy and physically active male subjects

Exclusion Criteria:

* Subjects who have latex allergy, hypertension, venous thrombotic disease, cardio-respiratory disease, or neurological disorders, acute and or chronic neuromuscular injuries i.e., with a history of serious lower limb injuries in 12 months period prior to study began will be excluded.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only male subjects will be recruited
Enrollment: 19 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Tensiomyography | 20 seconds per single measurement
  We will use TMG to assess PAP from pre to post-different tissue flossing procedures. The contractile properties of the individual muscles will be assessed by the non-invasive TMG method. We will measure the vastus lateralis muscle of the dominant leg only.
Countermovement jump | 30 seconds per single measurement
  Countermovement and squat jumps will be used to assess muscle fatigue from pre to post-different Vo2max testing procedures. Jumping ability will be assessed by vertical jump tests, using a bilateral force plate (model 9260AA6, Kistler, Switzerland) with Kistler MARS software to record ground reaction force data.

SECONDARY OUTCOMES:
Rate of perceived exertion | 5 seconds
  Rate of perceived exertion will be measured to assess subjective perception of the fatigue from pre-to post flossing procedure

CONTACTS AND LOCATIONS:
Overall Officials: Armin Paravlic, PhD, Principal Investigator — Faculty of Sport
Locations (1):
- Faculty of Sport, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No
We can share our data upon a reasonable request to the principal investigator

REFERENCES:
- [Result] Paravlic AH, Segula J, Drole K, Hadzic V, Pajek M, Vodicar J. Tissue Flossing Around the Thigh Does Not Provide Acute Enhancement of Neuromuscular Function. Front Physiol. 2022 Apr 27;13:870498. doi: 10.3389/fphys.2022.870498. eCollection 2022. PMID 35574482
- See also: Publisher site — https://www.frontiersin.org/articles/10.3389/fphys.2022.870498/full